CLINICAL TRIAL: NCT01482429
Title: Implantation of a Multidisciplinary Ventilator-weaning Protocol in a Intensive Care Unit of Teaching Hospital of Federal University of Uberlandia
Brief Title: Evaluation of a Systematic Approach to Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Liliane Barbosa da Silva Passos, Principal Investigator, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Desmame
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Weaning Failure; Complication of Respirator [Ventilator]
Keywords: ventilator weaning; protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protocol-directed (Experimental): Discontinuation of ventilation was based in multidisciplinary protocol.
  Interventions: Other: Multidisciplinary weaning-ventilator protocol
- Usual care (No Intervention): Discontinuation of ventilation was left entirely to the discretion of the physicians.

INTERVENTIONS:
Other: Multidisciplinary weaning-ventilator protocol — We implemented a multidisciplinary protocol for weaning from mechanical ventilation.This consist of a daily screening for readiness, performing a spontaneous breathing test, evaluation of signs of intolerance and decision on extubation.
  Other Names: Weaning-ventilator protocol
  Arms: Protocol-directed

SUMMARY:
Prolongation of mechanical ventilation poses serious personal and financial threats to healthcare consumers.

The investigators objectives are create and implement an multidisciplinary evidenced-based ventilator-weaning protocol to assess whether a systematic approach compared with the physician's judgment only decreases time spent on the ventilator, complications of mechanical ventilation and length of stay in critical care unit.

ELIGIBILITY:
Inclusion Criteria:

* remain in mechanical ventilation for more than 24 hours
* begin weaning from mechanical ventilation

Exclusion Criteria:

* admitted in the unit already in weaning from mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliane Barbosa da Silva Passos, Principal Investigator — Federal University of Uberlandia; Thulio Marquez Cunha, Study Chair — Federal University of Uberlandia; Carlos Henrique Alves de Rezende, MD, Study Chair — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients hospitalized in the intensive care unit, remained on mechanical ventilation for more than 24 hours and subjected to weaning from mechanical ventilation.
Period: Care Usual
Arm/Group | Protocol-directed | Usual Care
Started | 0 | 269
Completed | 0 | 96
Not Completed | 0 | 173
Not completed — Protocol Violation | 0 | 172
Not completed — Lost to Follow-up | 0 | 1
Period: Protocol
Arm/Group | Protocol-directed | Usual Care
Started | 414 | 0
Completed | 139 | 0
Not Completed | 275 | 0
Not completed — Protocol Violation | 275 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocol-directed | Usual Care | Total
Number analyzed (Participants) | 139 | 96 | 235
Age Continuous [Mean (Standard Deviation); unit: years] | 49.9 (20.18) | 43.5 (17.89) | 47.28 (19.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 101 | 63 | 164
Region of Enrollment [Number; unit: participants]
  Brazil | 139 | 96 | 235

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: length of ICU stay (days)
Population: Overall
Measure: Number; unit: participants
Arm/Group | Protocol-directed | Usual Care
Number analyzed (Participants) | 139 | 96
participants | 10 | 14
Statistical Analysis 1: Comparison: Protocol-directed vs Usual Care; Test type: Superiority or Other; p = 0.03, binomial test

2. Primary Outcome: Duration of Weaning From Mechanical Ventilation
Time Frame: days
Population: overall
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Protocol-directed | Usual Care
Number analyzed (Participants) | 139 | 96
days | 3.6 (5.49) | 6.8 (9.45)
Statistical Analysis 1: Comparison: Protocol-directed vs Usual Care; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Duration of Mechanical Ventilation
Time Frame: days
Reporting Status: Not Posted

4. Primary Outcome: Length of Intensive Care Unit Stay
Time Frame: days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Protocol-directed | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The lack of sedation protocol in the intensive care unit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No